CLINICAL TRIAL: NCT05704608
Title: Effects of an Aerobic Training Program on Liver Functions in Male Athletes - a Randomized Controlled Trial
Brief Title: Effects of Aerobic Training Program On Liver Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Masood Khan, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: DN 4900 /FSS
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Liver Functions
Keywords: Fatty liver; Physical activity; Treadmill; Exercises
MeSH Terms: conditions — Fatty Liver; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Aerobic training program was performed by participants.
  Interventions: Other: Aerobic training
- Control group (No Intervention): No intervention was performed by the participants.

INTERVENTIONS:
Other: Aerobic training — Exercises on a treadmill at different speeds and inclination were performed.
  Arms: Experimental Group

SUMMARY:
The liver plays a central role in energy exchange, protein synthesis as well as the elimination of waste products from the body. The optimal functioning of the liver is essential for athletic performance. It becomes necessary to maintain the enzymes of the liver at an optimal level so that liver cells can be protected from inflammation or damage. This paper investigated the effects of a twelve-week aerobic exercise program on the liver function of adult athletes. A total of thirty (30) healthy male athletes aged 21 to 24 were recruited for this study and kept in two equal groups. The control group was kept under rigorous supervision and did not participate in any special activities. The experiment group was well-versed in their assigned training program and solely performed the experimental procedure for twelve (12) weeks. Evaluation of all patients in both experimental and control groups was carried out before and after the treatment program by measuring the levels of (Alkaline phosphate, AST/SGOT, ALT/SGPT, Bilirubin Total/indirect/direct, Albumin, Globulin, and Total protein) respectively using standard methods by collecting blood samples, 5 mls each of baseline into lithium heparin containers for estimation of above biochemical parameters at the pathology laboratory accredited by National Accreditation Board for Testing and Calibration Laboratories accredited (NABL, India).

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age: 21-24 years
* Healthy
* Athletes

Exclusion Criteria:

* history of severe illness,
* surgery, or damage to liver,
* fatty liver disease,
* cirrhosis,
* blood infections,
* neuromuscular illnesses,
* or the presence of any disorders such as fever, high blood pressure, high blood sugar

Ages: 21 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Bilirubin-Total | 12 weeks.
  Blood level of Bilirubin-Total was measured.
Serum aspartate aminotransferase/serum glutamic-oxaloacetic transaminase (AST/SGOT) | 12 weeks.
  Blood level of Serum AST/SGOT was measured.
Serum alanine transaminase/Serum Glutamic Pyruvic Transaminase (ALT/SGPT) | 12 weeks.
  Blood level of Serum ALT/SGPT was measured.
Alkaline Phosphatase | 12 weeks.
  Blood level of Alkaline Phosphatase was measured.
Protein-Total | 12 weeks.
  Blood level of Protein-Total was measured.
Albumin | 12 weeks.
  Blood level of Albumin was measured.
Globulin | 12 weeks.
  Blood level of Globulin was measured.

CONTACTS AND LOCATIONS:
Overall Officials: Masood Khan, M.P.Th, Principal Investigator — King Saud University
Locations (1):
- King Saud University, Riyadh, Saudi Arabia